CLINICAL TRIAL: NCT06849921
Title: Precise Design of Cell Therapy for Relapsed and Refractory Hematological Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, MD, Ruijin Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ruijinH-KY2024-394
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-11

CONDITIONS: Precise Design of Cell Therapy for Relapsed and Refractory Hematological Tumors; Hematologic Disease
Keywords: cell therapy; hematological tumors
MeSH Terms: conditions — Hematologic Neoplasms; Hematologic Diseases | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Precise Design of CAR-cell Injection (Experimental): The drug for this trial is Precise Designof CAR- cells transduced with the lentiviral vector . The dose is 2x10e6 ~1x10e7 CAR-cell/kg in patients with relapsed/refractory hematologic malignancies.
  Interventions: Drug: Cellular Therapy

INTERVENTIONS:
Drug: Cellular Therapy — This intervention involves the infusion of autologous or allogeneic CAR-T cells into patients with relapsed/refractory hematologic malignancies. CAR-T cells are modified to target specific antigens on the surface of cancerous cells. After the infusion, patients will be monitored for response and safety.
  Administration: Intravenous infusion. Dosage: The maximum tolerated dose (MTD) will be determined as part of the study, with dose escalation used to identify the optimal and safest dose of CAR-T cells for treatment.

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of CAR-T cell therapy in patients with relapsed/refractory hematologic malignancies.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the efficacy and safety of CAR-T cell therapy in patients with relapsed/refractory hematologic malignancies. The primary objective is to determine the maximum tolerated dose (MTD), safety profile, and the overall response rate (ORR) of CAR-T cells in these patients. Secondary objectives include assessing marrow remission rates and minimal residual disease (MRD) clearance at various time points (2 weeks, 1 month, 3 months, 6 months, and 1 year) in patients with bone marrow involvement, as well as evaluating the changes in multiple sites of involvement through PET-CT or PET-MRI before and one year after CAR-T therapy. The study will also track event-free survival (EFS), progression-free survival (PFS), and overall survival (OS) rates at 1, 2, 3, and 5 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with relapsed/refractory hematologic malignancies confirmed to express CD19, CD22, CD20, CD7, CD5, CD2, CD79b, BCMA, GPCR5D, CD38, CD33, CD123, CD133, CLL1, EBV (GP350, LMP1), CMV (Gb21, gB280…) or other validated targets (supported by domestic and international preclinical/clinical evidence) who meet the following criteria:

Male or female, aged ≥18 years and <75 years; Newly diagnosed patients with refractory disease (as defined by respective diagnostic criteria) after chemotherapy; Newly diagnosed patients with disease progression during chemotherapy and poor anticipated response to further chemotherapy; Patients with relapsed disease (≥1 recurrence) and confirmed residual tumor evidence; Patients with relapse after autologous or allogeneic hematopoietic stem cell transplantation (HSCT); Patients with relapse after CAR-T therapy; Patients with hematologic malignancies deemed incurable by current surgical, radiotherapy, or chemotherapy interventions.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded:

Life expectancy <12 weeks; Genetic testing reveals mutations or structural variants associated with the target antigens; Severe graft-versus-host disease (GVHD) requiring immunosuppressive therapy in post-HSCT relapse patients; Post-HSCT relapse <3 months with no available donor;

Organ dysfunction:

Serum creatinine >2.5 mg/dL; ALT/AST >5× upper limit of normal (ULN); Total bilirubin >2 mg/dL; Uncontrolled active infection; Active hepatitis B/C or HIV infection; Anticipated early loss to follow-up (<3 months post-treatment); Failure to provide signed informed consent or lack of ethics committee approval; Concurrent systemic conditions that may interfere with study participation; Other exclusion criteria deemed appropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
adverse events. | 1 month
  Type, incidence and severity of adverse events
Maximum tolerated dose | 1 month
  The maximum dose that does not cause death of the subject
Overall response rate | 3 months
  ORR in patients is defined as the rate of complete remission (CR, CRh)

SECONDARY OUTCOMES:
Overall incidence and severity of adverse events. | 12 months
  Overall incidence and severity of adverse events will measure in this trial.
Rate of relapse and refractory of Hematologic Diseases patients achieving MRD negative CR | 12 months
  The rate of relapse and refractory of Hematologic Diseases patients achieving MRD negative CR in D28; 3,6,12months.

OTHER OUTCOMES:
Level of circulating CAR T cells | 12 months
  To investigate the relationship between the dynamic changes of CAR-T cells in the peripheral blood and treatment outcomes, as detected by FCM and/or real-time quantitative PCR technology

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No